CLINICAL TRIAL: NCT03226561
Title: Assessment of Near Vision Capacity in Different Light Conditions Following Bilateral Trifocal Intraocular Implantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Associate Professor, Democritus University of Thrace
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 334/20-7-2017
Record Dates: First submitted 2017-07-20; First posted 2017-07-24 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Panoptix Group (Active Comparator): Patients will receive bilateral phacoemulsification with diffractive trifocal lenses implantation (Phaco / Panoptix)
  Interventions: Procedure: Phaco / Panoptix
- Control Group (No Intervention): Control, age-matched presbyopic group corrected with presbyopic glasses

INTERVENTIONS:
Procedure: Phaco / Panoptix — Phacoemulsification with bilateral diffractive trifocal lens implantation
  Arms: Panoptix Group

SUMMARY:
Patients who underwent presbyopic correction with bilateral trifocal intraocular lenses implantation are supposed to have sufficient uncorrected vision capacity for activities of daily living (ADLs) that require near vision acuity (NV), (ie. book reading). However, it is known that light intensity and temperature has a great impact on near vision capacity. Primary objective of this study is to identify the optimal task lighting conditions (in terms of light intensity and temperature) for ADLs that demand near vision acuity for a sample of patients who underwent presbyopic correction with bilateral trifocal intraocular lenses implantation

DETAILED DESCRIPTION:
Patients who underwent presbyopic correction with bilateral trifocal intraocular lenses implantation are supposed to have sufficient uncorrected vision capacity for activities of daily living (ADLs) that require near vision acuity (NV), (ie. book reading). However, it is known that light intensity and temperature has a great impact on near vision capacity. Primary objective of this study is to identify the optimal task lighting conditions (in terms of light intensity and temperature) for ADLs that demand near vision acuity for a sample of patients who underwent presbyopic correction with bilateral trifocal intraocular lenses implantation. The following light intensities will be evaluated: 25, 50, and 75 foot candles. Moreover, the following light temperatures will be evaluated: 3000, 4000, and 6000 Kelvins.

ELIGIBILITY:
Inclusion Criteria:

Presbyopia

Exclusion Criteria:

Glaucoma Corneal pathology Fundus pathology Severe neurological/mental diseases that interfere with visual acuity

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
uNVC (3000K) | 6 months
  Uncorrected Near Vision Capacity at 3000 Kelvins
uNVC (4000K) | 6 months
  Uncorrected Near Vision Capacity at 4000 Kelvins
uNVC (6000K) | 6 months
  Uncorrected Near Vision Capacity at 6000 Kelvins
uNVC (25FC) | 6 months
  Uncorrected Near Vision Capacity at 25 Foot Candles
uNVC (50FC) | 6 months
  Uncorrected Near Vision Capacity at 50 Foot Candles
uNVC (75FC) | 6 months
  Uncorrected Near Vision Capacity at 75 Foot Candles

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD, PhD, Principal Investigator — Associate Professor
Locations (1):
- Democritus University of Thrace, Alexandroupoli, Evros, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Labiris G, Ntonti P, Panagiotopoulou EK, Konstantinidis A, Gkika M, Dardabounis D, Perente I, Sideroudi H. Impact of light conditions on reading ability following multifocal pseudophakic corrections. Clin Ophthalmol. 2018 Dec 14;12:2639-2646. doi: 10.2147/OPTH.S180766. eCollection 2018. PMID 30587911